CLINICAL TRIAL: NCT03402971
Title: Das Rechte Herz in Der Schwangerschaft. Echokardiographische Verlaufskontrollen Des Rechten Herzens während Und Nach Der Schwangerschaft.
Brief Title: The Right Heart During and After Pregnancy - an Echocardiographic Study
Acronym: EVA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gero Bunniger (Other)
Responsible Party: Sponsor-Investigator, Gero Bunniger, MD, University of Giessen
Organization: University of Giessen (Other)
Other Study IDs: 130/17
Record Dates: First submitted 2017-12-28; First posted 2018-01-18 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Pregnancy Related
Keywords: right heart; pregnancy; echocardiography; reference values
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy pregnant+healthy fetus: healthy pregnant women with suspected healthy fetus will get one echocardiography examination each trimester of pregnancy and one after delivery
  Interventions: Diagnostic Test: echocardiography
- non healthy pregnant: non healthy women with suspected healthy or unhealthy fetus will get one echocardiography examination each trimester of pregnancy and one after delivery
  Interventions: Diagnostic Test: echocardiography
- non healthy fetus: healthy or non healthy pregnant women with suspected non healthy fetus will get one echocardiography examination each trimester of pregnancy and one after delivery
  Interventions: Diagnostic Test: echocardiography

INTERVENTIONS:
Diagnostic Test: echocardiography — echocardiography focused on right heart: Parameters include RV enddiastolic diameter basal, mid-cavity and longitudinal, RVOT distal, pulmonal outflow AT and AT/ET, endsystolic RA area. RV wall thickness, TAPSE, S', tricuspidal E/A, E/e', RIMP. V. Cava to estimate CVP and sPAP.
  Other Names: parallel EKG

SUMMARY:
The main goal is to establish echocardiographic reference values of the right heart for pregnant women, assuming they differ significantly from those of non pregnant women of same age.

Therefore the investigators will use existing reference values published by American society of echocardiography and European Association of Echocardiography. As side arms the investigators want to explore, whether illness of either fetus or mother is connected with right heart affection.

DETAILED DESCRIPTION:
A lot of lung diseases affect the heart, too - especially the right heart. Well known examples are pulmonary embolism or pulmonary hypertension. But rather unknown is the fact, that right heart function presents as a prognostic parameter in a lot of (left heart) diseases, for example myocardial infarction, atrial fibrillation, left heart failure, but also in chronic obstructive pulmonary disease (COPD) or may be even diabetes mellitus. Since the left part of the heart has been studied by researchers more than fifty years, the right heart has moved into scientific focus not long ago.

The tool of choice to examine the living heart is echocardiography. There are no relevant risks or complications.

During an echocardiographic examination a lot of parameters are collected. To judge data in a clinical way reference values belonging to healthy persons are essential. Those values are highly dependant on sex, body size, age etc.

Since pregnancy changes a lot in the human body, reference values from non pregnant woman of same age (published by American society of echocardiography and European Association of Echocardiography) are presumably not representative. So the investigators want to establish echocardiographic reference values of the right heart for pregnant women. Therefore an echocardiographic examination will be applied within each trimester of pregnancy and after delivery. As side arms the investigators want to explore, whether illness of either fetus or mother is connected with right heart affection.

ELIGIBILITY:
Inclusion Criteria:

* pregnant
* 18years or older

Exclusion Criteria:

* acute illness demanding instant therapy
* poor or none sonographic results

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: women over 18 years, actual mean age is 33y
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-11-02 (Actual); Primary Completion 2023-11-02 (Estimated); Study Completion 2024-11-02 (Estimated)

PRIMARY OUTCOMES:
change in right ventricular (RV) enddiastolic diameter basal | first examination within 1st to 12th week of pregnancy, second examination within 13th to 28th week of pregnancy, third examination after 28th week of pregnancy and before delivery, fourth examination will take place at least 14 days after delivery
  The investigators measure right ventricular (RV) enddiastolic diameter basal (unit: mm), via echocardiography in apical 4 Chamber view, EKG-controlled.
change in RV enddiastolic diameter mid-cavitiy | first examination within 1st to 12th week of pregnancy, second examination within 13th to 28th week of pregnancy, third examination after 28th week of pregnancy and before delivery, fourth examination will take place at least 14 days after delivery
  The investigators measure right ventricular RV enddiastolic diameter mid-cavity (unit: mm), via echocardiography in apical 4 Chamber view, EKG-controlled.
change in RV enddiastolic diameter longitudinal | first examination within 1st to 12th week of pregnancy, second examination within 13th to 28th week of pregnancy, third examination after 28th week of pregnancy and before delivery, fourth examination will take place at least 14 days after delivery
  The investigators measure right ventricular RV enddiastolic diameter longitudinal (unit: mm), via echocardiography in apical 4 Chamber view, EKG-controlled.
change in right ventricular outflow tract (RVOT) distal | first examination within 1st to 12th week of pregnancy, second examination within 13th to 28th week of pregnancy, third examination after 28th week of pregnancy and before delivery, fourth examination will take place at least 14 days after delivery
  The investigators measure RVOT distal (unit: mm), via echocardiography in parasternal short-axis view, EKG-controlled.
change in right atrial (RA) endsystolic area | first examination within 1st to 12th week of pregnancy, second examination within 13th to 28th week of pregnancy, third examination after 28th week of pregnancy and before delivery, fourth examination will take place at least 14 days after delivery
  The investigators measure RA endsystolic area (unit: cm²), via echocardiography in apical 4 Chamber view, EKG-controlled.
change in RV wall thickness | first examination within 1st to 12th week of pregnancy, second examination within 13th to 28th week of pregnancy, third examination after 28th week of pregnancy and before delivery, fourth examination will take place at least 14 days after delivery
  The investigators measure RV wall thickness (unit: mm), via echocardiography in subcostal view, EKG-controlled. RV wall >5mm indicates RV hypertrophy.
change in tricuspid annular plane systolic excursion (TAPSE) | first examination within 1st to 12th week of pregnancy, second examination within 13th to 28th week of pregnancy, third examination after 28th week of pregnancy and before delivery, fourth examination will take place at least 14 days after delivery
  The investigators measure TAPSE (unit: mm), via echocardiography in apical 4 Chamber view + M-Mode at lateral tricuspid annulus, EKG-controlled. TAPSE is a parameter describing systolic RV-function.
change in S' velocity | first examination within 1st to 12th week of pregnancy, second examination within 13th to 28th week of pregnancy, third examination after 28th week of pregnancy and before delivery, fourth examination will take place at least 14 days after delivery
  The investigators measure S' velocity (unit: cm/sec), via echocardiography in apical 4 Chamber view + pulsed tissue Doppler velocity of the lateral tricuspid annulus, EKG-controlled. S' is a parameter describing systolic RV-function.
change in tricuspid E/A ratio | first examination within 1st to 12th week of pregnancy, second examination within 13th to 28th week of pregnancy, third examination after 28th week of pregnancy and before delivery, fourth examination will take place at least 14 days after delivery
  The investigators measure tricuspidal E/A ratio (unit: no unit), via echocardiography in apical 4 Chamber view + pulsed wave doppler over tricuspid inflow, EKG-controlled. Tricuspid E/A ratio is a parameter describing diastolic RV-function.
change in tricuspid E/e' ratio | first examination within 1st to 12th week of pregnancy, second examination within 13th to 28th week of pregnancy, third examination after 28th week of pregnancy and before delivery, fourth examination will take place at least 14 days after delivery
  The investigators measure tricuspid E/e' ratio (unit: no unit), via echocardiography in apical 4 Chamber view + pulsed wave doppler over tricuspid inflow + pulsed tissue Doppler velocity of the lateral tricuspid annulus, EKG-controlled. Tricuspid E/e' ratio is a parameter describing diastolic RV-function.
change in right index of myocardial performance (RIMP) | first examination within 1st to 12th week of pregnancy, second examination within 13th to 28th week of pregnancy, third examination after 28th week of pregnancy and before delivery, fourth examination will take place at least 14 days after delivery
  The investigators measure RIMP (unit: no unit), via echocardiography in apical 4 Chamber view + pulsed tissue Doppler velocity of the lateral tricuspid annulus, EKG-controlled. RIMP is calculated (isovolumic contraction time + isovolumic relaxation time) devided by (ejection time). RIMP is a parameter describing systolic RV-function.
change in inferior vena cava (IVC) diameter at end-expiration | first examination within 1st to 12th week of pregnancy, second examination within 13th to 28th week of pregnancy, third examination after 28th week of pregnancy and before delivery, fourth examination will take place at least 14 days after delivery
  The investigators measure IVC (unit: mm) via echocardiography subcostal or IVC view at end-expiration. IVC diameter correlates with central venous pressure.
change in inferior vena cava (IVC) diameter with sniff test. | first examination within 1st to 12th week of pregnancy, second examination within 13th to 28th week of pregnancy, third examination after 28th week of pregnancy and before delivery, fourth examination will take place at least 14 days after delivery
  The investigators measure IVC (unit: mm) via echocardiography subcostal or IVC view at forced inspiration. IVC diameter correlates with central venous pressure.
change in tricuspid regurgitation peak velocity | first examination within 1st to 12th week of pregnancy, second examination within 13th to 28th week of pregnancy, third examination after 28th week of pregnancy and before delivery, fourth examination will take place at least 14 days after delivery
  The investigators measure tricuspid regurgitation peak velocity (unit: m/sec) via echocardiography in apical 4 Chamber view + continuous wave doppler over tricuspid inflow respectively tricuspid regurgitation, if there is a tricuspid insufficiency, EKG-controlled. Tricuspid regurgitation peak velocity correlates with systolic pulmonary artery pressure (sPAP).
change in RV outflow tract acceleration time (RVOT-AT) | first examination within 1st to 12th week of pregnancy, second examination within 13th to 28th week of pregnancy, third examination after 28th week of pregnancy and before delivery, fourth examination will take place at least 14 days after delivery
  The investigators measure RVOT-AT (unit: msec) via echocardiography in parasternal short-axis view + pulsed wave doppler over pulmonal valve, EKG-controlled. RVOT-AT correlates with systolic pulmonary artery pressure (sPAP).

CONTACTS AND LOCATIONS:
Overall Officials: Henning Gall, Prof., MD, Principal Investigator — Pulmology, Department of pulmonal Hypertension
Locations (1):
- University of Gießen, Giessen, Hesse, Germany